CLINICAL TRIAL: NCT02044991
Title: The Efficacy of Ultrasound Guided Posterior Sacroiliac Ligament Corticosteroid Injection in Pregnancy-Related Pelvic Girdle Pain: A Randomized Controlled Trial
Brief Title: Ultrasound Guided Posterior Sacroiliac Ligament Corticosteroid Injection in Pregnancy-Related Pelvic Girdle Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted prematurely due to poor recruitment
Sponsor: Loyola University (Other)
Collaborators: American Academy of Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Colleen Fitzgerald, M.D., Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205418
Record Dates: First submitted 2014-01-17; First posted 2014-01-24 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Pelvic Girdle Pain
Keywords: Sciatica; Pelvic girdle pain
MeSH Terms: conditions — Pelvic Girdle Pain; Sciatica | interventions — Adrenal Cortex Hormones; Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive either an injection of methylprednisolone acetate plus lidocaine or to receive an injection of saline with lidocaine using a randomized block design with a 1:1 allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Participants randomized to this arm will receive a corticosteroid. This is 40mg of a non-fluorinated injectable glucocorticoid, methylprednisolone acetate (1cc) combined with 1cc of 1% Lidocaine
  Interventions: Drug: Corticosteroid
- Placebo (Placebo Comparator): Participant's randomized to this condition will receive a placebo injection once weekly
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: Corticosteroid — 40mg of a non-fluorinated injectable glucocorticoid, methylprednisolone acetate (1cc) combined with 1cc of 1% Lidocaine
  Other Names: Medrol
  Arms: Treatment
Drug: Placebo Injection — A placebo injection
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if pelvic girdle pain can be more effectively treated with the use of injectable anti-inflammatory medication plus physical therapy compared with physical therapy and a saline injection.

DETAILED DESCRIPTION:
Pelvic girdle pain (PGP) in pregnancy is common with prevalence estimates of 45%.1 It is defined as pain experienced between the posterior iliac crest and the gluteal fold, particularly in the region of the sacroiliac joint.2 Pain may radiate in the posterior thigh and can also occur in conjunction with/or separately in the symphysis. In PGP, the endurance capacity for standing, walking and sitting is diminished. The diagnosis of PGP can be reached after exclusion of lumbar causes and must be reproducible by specific clinical tests. While various pain mechanisms including mechanical, hormonal, inflammatory, and neural have been proposed in the development of PGP, the etiology and pathogenesis is poorly understood. It is possible that musculoskeletal changes influenced by hormonal (Relaxin) elevation in pregnancy predispose pregnant women to acute musculoskeletal injury presenting clinically as PGP. An inflammatory response in other acute musculoskeletal injuries has been well described3 and may also occur in pregnancy related PGP particularly given the musculoskeletal vulnerability during this time. Though PGP is common in pregnancy, no study to date has investigated the efficacy of anti-inflammatory treatment in pregnancy related PGP in order to better establish the contribution of inflammation in the etiology of pregnancy related PGP.

ELIGIBILITY:
Inclusion Criteria:

* Women who are not doing other therapies for pain (physical therapy, chiropractic management, pool)
* Women between age 21 and 50 who plan to deliver at Loyola or Gottlieb
* Pain Numeric Rating Scale (NRS) on average of greater than or equal to 5/10 at Visit 1
* Pain must be between the upper level of the iliac crests and the gluteal folds in conjunction with or separately from pain in the pubic symphysis and influenced by position and locomotion
* 2/4 positive physical examination tests on the symptomatic side including the P4 test, the LDL test, pubic symphysis palpation and the acute straight leg rise (ASLR)

Exclusion Criteria:

* Women presenting with PGP in the first or third trimester (<13 weeks gestation or >28 weeks gestation)
* Women with pubic symphysis (anterior) pain alone
* Women who do not plan to deliver a baby at Loyola or Gottlieb
* Pain above the upper level of the iliac crest
* History of lumbar or pelvic fracture, neoplasm, inflammatory disease, active urogenital infection or active gastrointestinal illness, current physical therapy or other therapies for PGP, or previous surgery of the lumbar spine, pelvic girdle, hip joint or femur
* History or signs of radiculopathy or other systemic neurologic disease
* Women with diabetes or gestational diabetes

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Fitzgerald, MD, Principal Investigator — Loyola Univ Med Cntr-
Locations (1):
- Loyola University Health System, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Wu WH, Meijer OG, Uegaki K, Mens JM, van Dieen JH, Wuisman PI, Ostgaard HC. Pregnancy-related pelvic girdle pain (PPP), I: Terminology, clinical presentation, and prevalence. Eur Spine J. 2004 Nov;13(7):575-89. doi: 10.1007/s00586-003-0615-y. Epub 2004 Aug 27. PMID 15338362
- [Background] Ekman EF, Koman LA. Acute pain following musculoskeletal injuries and orthopaedic surgery: mechanisms and management. Instr Course Lect. 2005;54:21-33. PMID 15948432
- [Background] Kristiansson P, Svardsudd K, von Schoultz B. Serum relaxin, symphyseal pain, and back pain during pregnancy. Am J Obstet Gynecol. 1996 Nov;175(5):1342-7. doi: 10.1016/s0002-9378(96)70052-2. PMID 8942512
- [Background] Stapleton DB, MacLennan AH, Kristiansson P. The prevalence of recalled low back pain during and after pregnancy: a South Australian population survey. Aust N Z J Obstet Gynaecol. 2002 Nov;42(5):482-5. doi: 10.1111/j.0004-8666.2002.00482.x. PMID 12495090
- [Background] Gutke A, Josefsson A, Oberg B. Pelvic girdle pain and lumbar pain in relation to postpartum depressive symptoms. Spine (Phila Pa 1976). 2007 Jun 1;32(13):1430-6. doi: 10.1097/BRS.0b013e318060a673. PMID 17545912
- [Background] Brynhildsen J, Hansson A, Persson A, Hammar M. Follow-up of patients with low back pain during pregnancy. Obstet Gynecol. 1998 Feb;91(2):182-6. doi: 10.1016/s0029-7844(97)00630-3. PMID 9469272
- [Background] Stuge B, Hilde G, Vollestad N. Physical therapy for pregnancy-related low back and pelvic pain: a systematic review. Acta Obstet Gynecol Scand. 2003 Nov;82(11):983-90. doi: 10.1034/j.1600-0412.2003.00125.x. PMID 14616270
- [Background] Stuge B, Laerum E, Kirkesola G, Vollestad N. The efficacy of a treatment program focusing on specific stabilizing exercises for pelvic girdle pain after pregnancy: a randomized controlled trial. Spine (Phila Pa 1976). 2004 Feb 15;29(4):351-9. doi: 10.1097/01.brs.0000090827.16926.1d. PMID 15094530
- [Background] Albert H, Godskesen M, Westergaard J. Prognosis in four syndromes of pregnancy-related pelvic pain. Acta Obstet Gynecol Scand. 2001 Jun;80(6):505-10. PMID 11380285
- [Background] Stuge B, Veierod MB, Laerum E, Vollestad N. The efficacy of a treatment program focusing on specific stabilizing exercises for pelvic girdle pain after pregnancy: a two-year follow-up of a randomized clinical trial. Spine (Phila Pa 1976). 2004 May 15;29(10):E197-203. doi: 10.1097/00007632-200405150-00021. PMID 15131454
- [Background] Elden H, Fagevik-Olsen M, Ostgaard HC, Stener-Victorin E, Hagberg H. Acupuncture as an adjunct to standard treatment for pelvic girdle pain in pregnant women: randomised double-blinded controlled trial comparing acupuncture with non-penetrating sham acupuncture. BJOG. 2008 Dec;115(13):1655-68. doi: 10.1111/j.1471-0528.2008.01904.x. Epub 2008 Oct 15. PMID 18947338
- [Background] Haugland KS, Rasmussen S, Daltveit AK. Group intervention for women with pelvic girdle pain in pregnancy. A randomized controlled trial. Acta Obstet Gynecol Scand. 2006;85(11):1320-6. doi: 10.1080/00016340600780458. PMID 17091411
- [Background] Bastiaenen CH, de Bie RA, Wolters PM, Vlaeyen JW, Leffers P, Stelma F, Bastiaanssen JM, Essed GG, van den Brandt PA. Effectiveness of a tailor-made intervention for pregnancy-related pelvic girdle and/or low back pain after delivery: short-term results of a randomized clinical trial [ISRCTN08477490]. BMC Musculoskelet Disord. 2006 Feb 27;7:19. doi: 10.1186/1471-2474-7-19. PMID 16504165
- [Background] Lin J, Fessell DP, Jacobson JA, Weadock WJ, Hayes CW. An illustrated tutorial of musculoskeletal sonography: part I, introduction and general principles. AJR Am J Roentgenol. 2000 Sep;175(3):637-45. doi: 10.2214/ajr.175.3.1750637. No abstract available. PMID 10954443
- [Background] Le Goff B, Berthelot JM, Maugars Y. Ultrasound assessment of the posterior sacroiliac ligaments. Clin Exp Rheumatol. 2011 Nov-Dec;29(6):1014-7. Epub 2011 Dec 22. PMID 22206650
- [Background] Pekkafahli MZ, Kiralp MZ, Basekim CC, Silit E, Mutlu H, Ozturk E, Kizilkaya E, Dursun H. Sacroiliac joint injections performed with sonographic guidance. J Ultrasound Med. 2003 Jun;22(6):553-9. doi: 10.7863/jum.2003.22.6.553. PMID 12795552
- [Background] Schull WJ, Otake M. Cognitive function and prenatal exposure to ionizing radiation. Teratology. 1999 Apr;59(4):222-6. doi: 10.1002/(SICI)1096-9926(199904)59:43.0.CO;2-M. PMID 10331523
- [Background] Ruiz-Irastorza G, Khamashta MA. Managing lupus patients during pregnancy. Best Pract Res Clin Rheumatol. 2009 Aug;23(4):575-82. doi: 10.1016/j.berh.2009.04.004. PMID 19591786
- [Background] Baer AN, Witter FR, Petri M. Lupus and pregnancy. Obstet Gynecol Surv. 2011 Oct;66(10):639-53. doi: 10.1097/OGX.0b013e318239e1ee. PMID 22112525
- [Background] Roberts D, Dalziel S. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004454. doi: 10.1002/14651858.CD004454.pub2. PMID 16856047
- [Background] Ostensen M, Ramsey-Goldman R. Treatment of inflammatory rheumatic disorders in pregnancy: what are the safest treatment options? Drug Saf. 1998 Nov;19(5):389-410. doi: 10.2165/00002018-199819050-00006. PMID 9825952
- [Background] Cole BJ, Schumacher HR Jr. Injectable corticosteroids in modern practice. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):37-46. doi: 10.5435/00124635-200501000-00006. PMID 15712981
- [Background] Kumar N, Newman RJ. Complications of intra- and peri-articular steroid injections. Br J Gen Pract. 1999 Jun;49(443):465-6. PMID 10562748
- [Background] Slotkoff AT, Katz P. Approach to the patient with rheumatoid arthritis. Adv Intern Med. 1994;39:197-240. PMID 7908157
- [Background] Plastaras CT, Joshi AB, Garvan C, Chimes GP, Smeal W, Rittenberg J, Lento P, Stanos S, Fitzgerald C. Adverse events associated with fluoroscopically guided sacroiliac joint injections. PM R. 2012 Jul;4(7):473-8. doi: 10.1016/j.pmrj.2012.02.001. Epub 2012 Apr 28. PMID 22543036
- [Background] Jacobs JW, Michels-van Amelsfort JM. How to perform local soft-tissue glucocorticoid injections? Best Pract Res Clin Rheumatol. 2013 Apr;27(2):171-94. doi: 10.1016/j.berh.2013.03.003. PMID 23731930
- [Background] Elimian A, Goodman JR, Knudtson E, Wagner A, Wilson P, Williams M. Local anesthesia and pain perception during amniocentesis: a randomized double blind placebo-controlled trial. Prenat Diagn. 2013 Dec;33(12):1158-61. doi: 10.1002/pd.4214. Epub 2013 Sep 1. PMID 23939867
- [Background] Edelman A, Nichols MD, Leclair C, Astley S, Shy K, Jensen JT. Intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2004 Jun;103(6):1267-72. doi: 10.1097/01.AOG.0000127981.53911.0e. PMID 15172863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this trial began in May 2015 and ended in May 2016 (12 months). The trial was terminated in February 2017 due to poor recruitment
Groups:
- Treatment: Participants randomized to this arm receive an injectable anti-inflammatory medication (methylprednisolone acetate) plus lidocaine
- Placebo: Participant's randomized to this condition receive a saline injection with lidocaine.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all participants who signed an informed consent document to participate in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Pain is measured using the Pain Numeric Rating Scale (NRS), which ranges from 0 to 10 with higher scores indicating greater pain. This measure is recorded at baseline (0 weeks) and 8 weeks. The change in pain between these two time points (i.e., the difference score) is compared between the two groups.
Time Frame: 8 weeks
Population: The trial was prematurely terminated in February 2017 due to poor recruitment. No statistical analysis is conducted.
Measure: Median (Full Range); unit: change score on the NRS pain scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 2 | 0
change score on the NRS pain scale | -3 [-5 to -1] |

2. Secondary Outcome: Pelvic Functioning
Description: Pelvic functioning is measured at baseline (0 weeks) and week 8 using the Pelvic Girdle Questionnaire (PGQ), which ranges from 0 to 100 points with higher scores revealing greater pelvic girdle pain. The change in pelvic functioning between these two time points (i.e., the difference score) is compared between the two groups.
Time Frame: 8 weeks
Population: The trial was prematurely terminated in February 2017 due to poor recruitment. No statistical analysis is conducted.
Measure: Median (Full Range); unit: change score on the PGQ scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 2 | 0
change score on the PGQ scale | -35.5 [-75 to 4] |

3. Secondary Outcome: Disability
Description: Disability is measured at baseline (0 weeks) and week 8 using the Oswestry Disability Index (ODI), which is a measure of low back pain that ranges from 0 points to 100 with higher scores indicating greater disability. The change in disability between these two time points (i.e., the difference score) is compared between the two groups.
Time Frame: 8 weeks
Population: The trial was prematurely terminated in February 2017 due to poor recruitment. No statistical analysis is conducted.
Measure: Median (Full Range); unit: change score on the ODI scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 2 | 0
change score on the ODI scale | -15.25 [-44.5 to 14] |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year, 7 months
Description: For the placebo arm, the number of participants at risk for an adverse event, serious adverse event, and all-cause mortality is zero. This is because no participants were assigned to placebo. In this study, only two individuals were assigned to an intervention and both received the injectable anti-inflammatory medication (methylprednisolone acetate) plus lidocaine.
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=2) | Placebo (N=0)
Premature birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=2) | Placebo (N=0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Premature contractions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated in February 2017 due to poor recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02044991/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT02044991/ICF_001.pdf